CLINICAL TRIAL: NCT01832272
Title: The Effects of Tourniquet Reinflation After Early Tourniquet Release in Total Knee Arthroplasty
Brief Title: Reinflation After Early Tourniquet Release in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyun Kim, Direcor, Joint reconstruction center, SNUBH, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1206/158-004
Record Dates: First submitted 2013-02-20; First posted 2013-04-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Total knee arthroplasty; Tourniquet; Early release; Reinflation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reinflation after early deflation (Experimental): The tourniquet is released after cement implant fixation, and then reinflated, once arterial bleeding was controlled (Reinflation after early tourniquet deflation).
  Interventions: Procedure: Reinflation after early tourniquet deflation
- No reinflation after early deflation (No Intervention): The tourniquet is released after cement implant fixation, and remained deflated without reinflation, even after hemostasis.

INTERVENTIONS:
Procedure: Reinflation after early tourniquet deflation — The tourniquet is released after cement implant fixation, and then reinflated, once arterial bleeding was controlled
  Other Names: Reinflation after early tourniquet release
  Arms: Reinflation after early deflation

SUMMARY:
This study is aimed to determine the efficacy and the safety of the tourniquet reinflation after early tourniquet release in total knee arthroplasty, compared to the method of early deflation without reinflation. The investigators hypothesized that the reinflation after early release of the tourniquet would be effective in terms of improved visualization of the surgical field and decreased operation time and blood loss, whereas it would increase tourniquet-related complication due to longer tourniquet-use time.

DETAILED DESCRIPTION:
Total knee arthroplasty(TKA) is mostly performed with tourniquet applied, because it allows decreased intraoperative blood loss, better visualization of surgical field and better cement fixation of the implants, compared to the TKA without using tourniquet. However, there remains a controversy about the timing of tourniquet release, so the tourniquet may be unreleased throughout the whole operation time or released early just after cement fixation of the implants, atc. Early tourniquet release is generally aimed to control hidden arterial bleeding which would not be revealed if the tourniquet was unreleased. This method was reported to reduce arterial bleeding and its related complications, but it was also known that increase intraoperative bleeding, incidence of transfusion, and operation time. On the other hand, late tourniquet release, which the tourniquet is unreleased until the wound is closed, is reported to increase tourniquet-use time and related complications owing to longer tourniquet time, although it gives shorter operation time. The investigators have been used a way of reinflation of tourniquet after early release, once the arterial bleeding was controlled sufficiently, to balance the advantages and disadvantages of the early tourniquet release. The investigators were able to control arterial bleeding during the time the tourniquet was released, and the remained procedures were performed conveniently with good visualization of the surgical field after the tourniquet was reinflated again. However, there was no previous studies about the efficacy and the safety of the way of reinflation after early release of the tourniquet in the literature. Therefore, the investigators ask in this study whether the reinflation after early tourniquet release has advantages over the method of early tourniquet release without reinflation, in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis of the knee
* Scheduled for elective total knee arthroplasty
* Written signed consent

Exclusion Criteria:

* Revision TKA
* Diagnosis other than primary osteoarthritis
* Intra-articular indwelling drainage
* Refusing participate

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Operation time | from skin incision to wound closure
  Total time between initial skin incision and wound closure

SECONDARY OUTCOMES:
Tourniquet time | total sum of time between inflation and deflation of tourniquet
  Total time of tourniquet-use during the operation which defined from skin incision to the wound closure
Difficulty of the operation | from skin incision to wound closure
  Measured by the number of operative field clearance using gauze to make the remained procedure convenient
Incidence of transfusion | within 2weeks after surgery
  The incidence of allogenic or autologous (preoperative autologous blood donation) transfusion after surgery due to significant hemoglobin drop within 2weeks after surgery
Wound complications | on the 2nd and 14th day after surgery
  wound complications evaluated on the 2nd and 14th day after surgery, such as ecchymosis, subcutaneous hematoma, hemarthrosis, and oozing
Thigh complications | within 2 weeks
  Thigh complication due to the tourniquet, such as ecchymosis, skin bullae, and skin necrosis around the area of tourniquet application
Venous thromboembolism | within 2 weeks
  symptomatic deep vein thrombosis and pulmonary embolism, detected within 2weeks after surgery
Postoperative pain (VAS) | on the 2nd and 5th day after surgery.
  An independent investigator who was blinded to randomization assessed knee and thigh pain level using 0 to 10 visual analog scale (VAS) that ranged from 0 (no pain) to 10 (worst imaginable pain) on the 2nd and 5th day after surgery.
More painful site | on the 2nd and 5th day after surgery
  An independent investigator who was blinded to randomization assessed the more painful site either knee (operation site) or thigh (tourniquet application site) on the 2nd and 5th day after surgery.
More painful side in SBTKA | on the 2nd and 5th day after surgery.
  An independent investigator who was blinded to randomization assessed the more painful side in patients undergoing simultaneous bilateral TKA (SBTKA), whose each knee will be allocated into experimental and control group, respectively.
Amount of drainage | Until the drainage removal, average of 1 to 2 days after surgery
  Total amount of subcutaneous indwelled drainage before removal of it.
Hemoglobin drop on the 2nd day after surgery | On the 2nd day after surgery
  The hemoglobin drop calculated by subtracting hemoglobin level of postoperative 2nd day from the preoperative value
Hemoglobin drop on the 5th day after surgery | On the 5th day after surgery
  The hemoglobin drop calculated by subtracting hemoglobin level of postoperative 5th day from the preoperative value

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyun Kim, MD, PhD, Principal Investigator — Joint Reconstruction Center, Seoul National University Bundang Hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea